CLINICAL TRIAL: NCT06908395
Title: Impact of Everyday Light Exposure Patterns on Metabolic, Cardiovascular, and Psychological Health in Younger and Older Adults
Brief Title: Impact Of Everyday Light Exposure Patterns On Health
Acronym: AgeLight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Jan-Frieder Harmsen, Principal Investigator, RWTH Aachen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EK 24-324
Record Dates: First submitted 2025-03-20; First posted 2025-04-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Healthy Male and Female Subjects; Healthy Elderly
Keywords: Spectral diet; ambulatory assessment; daylight; m-path; eye degeneration; lense yellowing; continuous glucose monitoring; healthy aging; light sensitivity; melanopic EDI
MeSH Terms: conditions — Photophobia

STUDY DESIGN:
Intervention Model Description: This study is designed as an observatory field study of characterizing younger and older adults' everyday life over 10 days continuously through wearables and smartphone-based self-reports. In a randomized cross-over design, the 11th and 12th day will be spent in either bright (1250 lux) or dim office lighting (10 lux).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 days ambulatory assessment + 1 office day in bright light + 1 office day in dim light (Experimental): Day 11 is spent under laboratory conditions in bright (1250 lux) office lighting from 08:30 to 17:00 h. Day 12 is spent under laboratory conditions in dim (10 lux) office lighting from 08:30 to 17:00 h.
  Interventions: Other: 10-day ambulatory assessment in everyday life combined with two laboratory office days
- 10 days ambulatory assessment + 1 office day in dim light + 1 office day in bright light (Experimental): Day 11 is spent under laboratory conditions in dim (10 lux) office lighting from 08:30 to 17:00 h. Day 12 is spent under laboratory conditions in bright (1250 lux) office lighting from 08:30 to 17:00 h.
  Interventions: Other: 10-day ambulatory assessment in everyday life combined with two laboratory office days

INTERVENTIONS:
Other: 10-day ambulatory assessment in everyday life combined with two laboratory office days — Participants undergo a 10-day ambulatory assessment period wearing a continuous glucose monitor and a light logger as a necklace as well as completing short questionnaires through a smartphone app at regular intervals every day. On the first day, participants also undergo an extensive eye examination. Day 11 and 12 are spent in either dim or bright office lighting in randomized order.

SUMMARY:
The aim of the present study is to characterize everyday light conditions of younger and older adults and to consider them in relation to cardiovascular, metabolic and psychological health. An ambulatory assessment approach will be used over 12 days, measuring physiological parameters and daily thoughts, behaviors and experiences of different age groups using wearable technologies (e.g., light sensors, activity trackers, continuous glucose monitors) and smartphone-based self-reports (e.g., mood, vitality).

At the beginning of the study, the degeneration of the lens and retina of the participants is objectively quantified by ophthalmologists. On the last two days, participants will spend one working day in dim light and another in bright light in randomized order under the same measurement protocol as before in order to experimentally assess their sensitivity to light and its health effects.

DETAILED DESCRIPTION:
This study is designed as an observatory field study of characterizing younger and older adults' everyday life in terms of light exposure patterns as well as cardiovascular, metabolic and psychological health parameters over 10 days continuously through wearables and smartphone-based self-reports (ambulatory assessment period). On the first day of data collection, each participant will undergo an extensive eye examination at the Institute of Ophthalmology, particularly an Optical Coherence Tomography (OCT) scan will conducted and by means of a macular pigment reflectometer the difference between the light entering and leaving the eye across the visual spectrum will be determined as a marker of lense yellowing. Thereafter, participants start wearing the wearable sensors (continuous glucose monitors, light loggers worn as a necklace) and instructions on how to complete the smartphone-based self-report forms are provided. Participants are asked to take pictures of every food or drink (except of water) and upload these pictures through the m-Path app, these photos will be later linked to the continuous glucose monitor data. Data will be collected from the first evening onwards (ca. 18:00 h). After the ambulatory assessment period under free-living conditions, participants will spend the 11th and 12th day in a controlled office room environment from 08:30 to 17:00 h. In a randomized cross-over design, the 11th and 12th day will be spent in either bright (1250 lux) or dim office lighting (10 lux). On these days, participants will continue to wear the wearables and complete the expanded smartphone-based self-reports mostly similar to the 10-day ambulatory assessment period. Between day 11 and 12, participants will leave controlled conditions from 17:00 h on day 11 to 08:30 h on day 12. On day 11 and 12, participants will receive a standardized fluid meals for breakfast and lunch, and are otherwise instructed to avoid any food, caloric or caffeinated beverages between 08:30 and 17:00 h. On these two days, skin temperature sensors will be placed on four different skin regions, and blood pressure will be manually measured at regular intervals between 08:30 h and 17:00 h. After removing all wearables on day 12, the study ends at 17:30 h. Over these 12 days of data collection, participants will be asked to keep their bedtimes at home as consistent as possible between days, and on day 11 and 12 they will be instructed to come to the office facilities fasted without any caloric intake after 22:00 h on the previous evening of day 10 and 11, respectively.

The two comparative groups formed in this study consist of 30 younger adults (18-35 years) and 30 older adults (60-80 years), both females and males will be included, and the aim is to match both groups with respect to sex (i.e. ideally 15 women and 15 men per group). The age contrast in the two groups is chosen, as substantial differences in degeneration of the lenses and retina within the eye can be expected.

For the sample size calculation of n = 30 per group, we refer to Zauner et al. (Zauner et al., 2023), who created a procedure to calculate statistical power and required sample size for wearable light-logging data. For most light-logging metrics, their approach shows that for strong differences in light exposure patterns (i.e., winter vs. summer) even smaller samples are sufficient (n = 3-24). We do not expect that differences between age groups are that strong as seasonal differences. However, we are confident that effects of about d = 0.7 could be detected with our design (n = 30 per group). Considering some drop-out, we anticipate that we will have to enroll 70 participants in total.

With the primary hypothesis of this study being that younger and older individuals differ in their light exposure patterns in everyday life, the two main explorative goals of the AgeLight study are to:

* characterize light exposure patterns in younger and older adults and their link to cardiovascular, metabolic, and psychological health
* identify determining factors of an individual's sensitivity to light and its health effects (such as degeneration of the lens and retina)

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 or 60-80 years old
* Voluntary participation, signed consent form
* Owns an Android or iOS Smartphone compatible with the m-Path App
* Generally healthy (self-reported)
* Non-smoker for at least 12 months (self-reported)

Exclusion Criteria:

* Pregnancy (for female participants) (self-reported)
* Night-shift worker
* Eye diseases (e.g. glaucoma, age-related macular degeneration, diabetic retinopathy conditions after retinal detachment / retinal blood vessel occlusions)
* Pseudophakic eyes
* Psychological disorders: insomnia, depression, bipolar disorder and generalized anxiety disorder
* Wearing specially-filtered glasses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Mean melanopic EDI (lux) from 09:00 to 17:00 h (daytime in European winter months) | Over the 10-day ambulatory assessment period
  Measured via light loggers (ActLumus) worn as a necklace
Mean melanopic EDI (lux) 2 hours before individual bedtime | Over the 10-day ambulatory assessment period
  Measured via light loggers (ActLumus) worn as a necklace

SECONDARY OUTCOMES:
Lense degeneration | Baseline
  The macular pigment reflectometer will record the difference between the light entering and leaving the eye across the visual spectrum. Spectral analysis of the reflected light provides an adequate estimate of the yellowing of the intra-ocular lens.
Macular and retinal thickness | Baseline
  ophthalmologic evaluation of an Optical Coherence Tomography (OCT) scan
Interstitial glucose levels | Over the 10-day ambulatory assessment period, and specifically levels of day 11 and day 12 between 8:30 and 17:00 h upon controlled office lighting
  Interstitial glucose levels measured by continuous glucose monitors
Systolic and diastolic blood pressure | 09:00, 10:30, 12:00, 13:00, 14:30, 16:00 and 17:00 on day 11 and 12
  Manually measured via automated blood pressure cuffs
Heart rate | 09:00, 10:30, 12:00, 13:00, 14:30, 16:00 and 17:00 h on day 11 and 12
  Manually measured via automated blood pressure cuffs
Skin temperature | from 09:00 to 17:00 h on day 11 and 12
  in °C assessed via wireless temperature sensors (iButtons) placed on the hand, neck, clavicular and shin
Alertness | at least 6 times daily over all 12 study days
  measured via Karolinska Sleepiness Scale through the m-Path app
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  PSQI score calculated based on a digital questionnaire
Munich Chronotype Questionnaire (MCU) | Baseline
  Chronotype score calculated based on a digital questionnaire
Subjective sleep quality | every morning over the 12 study days
  measured via Consensus Sleep Diary through the m-Path app

OTHER OUTCOMES:
Digital food photo diary | continuously throughout the 12-day study period
  Participants take photos of every caffeine- or calorie-containing food item that they consume and upload them in the m-Path app

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Frieder Harmsen, PhD, Principal Investigator — RWTH Aachen University
Locations (1):
- University hospital at RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The study protocol can be requested via email to study officials.
Supporting Information: Study Protocol
Time Frame: The study protocol is available from the 20th of March 2025 onwards for at least 5 years.
Access Criteria: The study protocol can be requested via email to study officials.

DOCUMENTS (1):
  • Study Protocol (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT06908395/Prot_000.pdf